CLINICAL TRIAL: NCT05376956
Title: Comparison of Effect of Muscle Energy Technique vs PNF in Individuals With Hamstring Shortness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/505
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Hamstring Shortness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental): Using Muscle Energy Technique in Individuals With Hamstring Shortness
  Interventions: Diagnostic Test: Muscle Energy Technique
- Proprioception neuromuscular facilitation (PNF) (Experimental): Using proprioception neuromuscular facilitation (PNF) in Individuals With Hamstring Shortness
  Interventions: Diagnostic Test: Proprioception neuromuscular facilitation (PNF)

INTERVENTIONS:
Diagnostic Test: Muscle Energy Technique — Using Muscle Energy Technique in Individuals With Hamstring Shortness
  Arms: Muscle Energy Technique
Diagnostic Test: Proprioception neuromuscular facilitation (PNF) — Using proprioception neuromuscular facilitation (PNF) in Individuals With Hamstring Shortness
  Arms: Proprioception neuromuscular facilitation (PNF)

SUMMARY:
Comparison between the Effect of Muscle Energy Technique in Individuals with Hamstring Shortness and PNF in Individuals With Hamstring Shortness

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age group between 20 to 60 years with sedentary lifestyle will be included.
* both males and females will be included.
* Patients with diagnosed Tight hamstrings having knee extension less than 160º with the hip at 90º flexion.
* Patients with decreased ROM at the knee joint.
* Patients with reduced straight leg raise.
* Patients with pain in posterior compartment of thigh.
* Asymptomatic patients will be included.
* Patients with restricted mobility of lower limb due to Hamstring shortness.
* Symptomatic patients with hamstring tightness like of low back pain, pelvic tightness, knee osteoarthritis (grade 1 and 2) are included in the research.

Exclusion Criteria:

* Patients with prolapsed disc will excluded.(14)
* Patients with lower extremity injuries (strain, sprain, ligament injuries, etc.) in last 6 months will be excluded.
* Patients with severe hamstring injury either acute or chronic will be excluded.
* Patients with visual acute swelling in the region of hamstring muscle
* Patients with fracture of any type and area.
* Patients with dislocations or subluxations present will be excluded.
* Patient recommended for TKR of knee joint.
* Patients with any neurological disease like lumbar/cervical herniation, polyneuropathy, scoliosis etc.)
* Patient with any tumor of hip or knee with traumatic brain injury, spinal cord injuries will be excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Individuals With Hamstring Shortness | 6 Months
  Research will be effective to compare effectiveness of muscle energy technique MET and proprioceptive neuromuscular facilitation (PNF) to the further develop conclusion that which treatment method is more effective and quicker for the treatment of pain, improving flexibility and functional ability of patients with hamstring shortness having sedentary life style.
  Most of the target population having hamstring shortness due to sedentary lifestyle mostly poor posture and ergonomics that may eventually leads to loss of flexibility, functional ability and increases pain. The two procedures were applied at a very same time with equal gatherings and similar standards. Met and PNF are most effective stretching techniques to be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No